CLINICAL TRIAL: NCT03013738
Title: The Efficacy of the Growing Pro-Social (GPS) Program in Male Prison Inmates: A Randomized Controlled Trial
Brief Title: The Effects of the GPS Program in Offenders
Acronym: GPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Coimbra (Other)
Responsible Party: Principal Investigator, Nelio Brazao, MSc, University of Coimbra
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CINEICC-1-NB; SFRH/BD/89283/2012 (Other Grant/Funding Number: Portuguese Foundation for Science and Technology)
Record Dates: First submitted 2017-01-04; First posted 2017-01-06 (Estimated); Last update posted 2017-01-06 (Estimated); Status verified 2017-01

CONDITIONS: Male Prison Inmates
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Growing Pro-Social (GPS) program (Experimental): The Growing Pro-Social (GPS) program is a cognitive-behavioral group program for offenders. GPS is based on schema therapy, which conceptualizes aggressiveness as a result of a distorted view of the self and of the others. The ultimate goal of the GPS is to promote change in dysfunctional core beliefs about the self and the others.
  GPS consists of 40 sessions, each lasting about 90 minutes. Sessions must be carried out by two therapists who should be skillful in schema therapy. Sessions are grouped into five modules: (1) human communication, (2) interpersonal relationships, (3) cognitive distortions, (4) function and meaning of emotions, and (5) early maladaptive schemas.
  The treatment group attended the GPS program in addition to the Treatment AsUsual (TAU) delivered at Portuguese prisons.
  Interventions: Behavioral: Growing Pro-Social Program; Other: Treatment As Usual
- Treatment As Usual (Other): Subjects in this group received Treatment As Usual in Portuguese prisons (supervision of school frequency, occupational and job-related tasks and sentence planning supervision over time) and did not attend the GPS program or any other structured program during the research period.
  Interventions: Other: Treatment As Usual

INTERVENTIONS:
Behavioral: Growing Pro-Social Program — GPS is a structured cognitive-behavioral group program aimed to reduce the prominence of early maladaptive schemas
  Arms: Growing Pro-Social (GPS) program
Other: Treatment As Usual — TAU in Portuguese prisons is primarily aimed to increase educational and professional qualifications

SUMMARY:
This randomized controlled trial aimed to assess the efficacy of a 40-session cognitive-behavioral group program, Growing Pro-Social (GPS), in reducing early maladaptive schemas and cognitive distortions (primary outcomes), as well as anger, shame and paranoia (secondary outcomes). The GPS's impact on behavioral change (e.g., in the reduction of disciplinary incidents and prison records) was also tested, in order to ascertain if changes observed in cognitive and emotional variables were reflected in a more adjusted behavioral pattern. Personality Disorders were also tested as moderators of treatment effects.

DETAILED DESCRIPTION:
This was a randomized controlled trial with blind assessments, carried out in nine prisons in three city areas in mainland Portugal (Lisbon, Oporto and Coimbra) and in the Madeira Island.

After the study was approved by the Head of the General Directorate of Reintegration and Prison Services of the Portuguese Ministry of Justice, a list of potential participants who did not meet the exclusion criteria was made available to the research team by psychologists from the justice system. Next, a large sample of participants was randomly selected using a random number table by a research assistant who was blind to any personal information about each inmate. Then, a first meeting between the research team and the randomized inmates occurred, in which researchers invited inmates to participate voluntarily. In this meeting, researchers explained the goals of the study and presented a brief overview of the intervention program. It was also explained to inmates that their participation in the study would not impact their sentencing in any way.

Participants who agreed to participate, gave written informed consent, completed the baseline assessment, and were randomly assigned to treatment conditions (treatment and control groups) using a random number table by a research assistant who was blind to any information about each participant. Afterwards, the research team informed the psychologists in each prison of the result of the randomization so that GPS could be initiated. Participants in the control group were informed that they would be offered the GPS treatment after the study's completion (including the follow-up period).

Besides baseline assessment, participants completed the mid-assessment (after the 20th session of the program), post-treatment assessment (at the end of GPS) and follow-up assessment (12 months after GPS completion). Staff who conducted randomization did not serve as therapists or accessors, and accessors were blind to condition assignment. Respondent-specific codes were used to link the data from one time-point to the next one.

GPS's facilitators were chosen among the psychologists who already had training and experience in delivering the program with inmates (who were not selected for this study). In order to assure program integrity and consistency, facilitators received regular supervision by the research team (including the program's main author) during the time GPS was run in prisons. Moreover, the program's structured and manualized design ensures integrity, at least partially.

ELIGIBILITY:
Inclusion Criteria:

1. male prison inmates aged between 18 and 40 years old
2. remaining in prison for at least 24 months (taking into account GPS's 12-month length and 12-month follow-up assessment), since the beginning of the program.

Exclusion Criteria:

1. presence of cognitive disabilities (because GPS is not suitable for the cognitively-impaired)
2. psychotic symptoms (the experiential exercises used in the program are contraindicated for psychotic patients)
3. being treated for drug abuse/dependence (cessation or at least substantial reduction of drug or alcohol use must precede GPS treatment)
4. being sentenced exclusively for sexual offenses (sex offenders would benefit from more specific intervention programs)

NOTE: Female offenders were also excluded from the sample because women represent less than 6% of the total inmates in Portugal, and any possible idiosyncrasies from this cohort would be underrepresented.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 270 (Actual)
Dates: Start 2013-05; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Early maladaptive schemas | From baseline to 12 months' follow-up
  Participants reported on a questionnaire of early mal-adaptive schemas (EMSs), the Young Schema Questionnaire - YSQ-S3 (Young, 2005). The YSQ-S3 is a widely-used self-report questionnaire including 90 items, measuring the 18 EMSs proposed by Young (1990). Each EMS is evaluated using a set of five items listed randomly, which the individual rates using a Likert-type scale from 1 (completely untrue to me) to 6 (describes me perfectly).
  This assessment was carried out by researchers, who received training in the self-report measure.
Cognitive distortions | From baseline to 12 months' follow-up
  Participants reported on a questionnaire of cognitive distortions, the Angry Cognitions Scale - ACS (Martin & Dahlen, 2007). The ACS consists of 54 items distributed across nine scenarios (e.g., "You get home from the drive-thru and realized that you were given the wrong food"). Participants are asked to imagine that the situation described in each scenario had just happened. For each scenario, there are six items referring to different thoughts that could arise during the situation, which can be rated on a five-point Likert-type scale (1 = very unlikely to 5 = very likely).
  This assessment was carried out by researchers, who received training in the self-report measure.

SECONDARY OUTCOMES:
Anger | From baseline to 12 months' follow-up
  Participants reported on a questionnaire of anger, the State-Trait Anger Expression Inventory - STAXI (Spielberger, 1988). The STAXI is a 44-item questionnaire divided into three parts: the first part assesses anger-state (how one feels in the present moment), the second part assesses anger-trait (how one generally feels), and the third part assesses anger-expression (how one generally reacts or behaves when feeling enraged or angry. Anger-trait encompasses two factors (temperament and angry-reaction), and anger-expression is composed by three factors (anger-in, anger-out and anger-control). Each item is rated on a four-point scale (1 = not at all to 4 = almost always).
  This assessment was carried out by researchers, who received training in the self-report measure.
External shame | From baseline to 12 months' follow-up
  Participants reported on a questionnaire of external shame, the Other as Shamer Scale - OAS (Allan, Gilbert, & Goss, 1994). The OAS is an 18-item scale that assesses external shame (i.e., subject's perception of being negatively judged by others). Each item is rated on a five-point scale (0 = never to 4 = almost always) according to how frequently the individual feels s/he is being judged by others (e.g., "Other people seem me as small and insignificant").
  This assessment was carried out by researchers, who received training in the self-report measure.
Paranoia | From baseline to 12 months' follow-up
  Participants reported on a questionnaire of paranoia, the Paranoia Scale - PS (Fenigstein & Vanable, 1992). The PS is a 20-item self-report measure that assesses paranoid ideation. Items are rated on a five-point Likert scale (1 = not at all applicable to 5 = extremely applicable), where higher scores suggest high paranoid ideation.
  This assessment was carried out by researchers, who received training in the self-report measure.
Emotion Regulation | From baseline to 12 months' follow-up
  Participants reported on a questionnaire of emotional regulation, the Emotion Regulation Questionnaire - ERQ (Gross & John, 2003). The ERQ is a 10-item scale designed to measure respondents' tendency to regulate their emotions in two ways: (1) Cognitive Reappraisal and (2) Expressive Suppression. Respondents answer each item on a 7-point Likert-type scale ranging from 1 (strongly disagree) to 7 (strongly agree).
  This assessment was carried out by researchers, who received training in the self-report measure.
Disciplinary incidents inside prison | From baseline to 12 months' follow-up
  For estimation of the frequency and type of disciplinary incidents and infractions, the individual records of each participant was collected from the prison records, describing their frequency and type during the research period.

OTHER OUTCOMES:
Personality Disorders | Baseline
  Participants were interviewed with the SCID-II - Structured Clinical Interview for DSM-IV Axis II Personality Disorders (First, Gibbon, Spitzer, Williams, & Benjamim, 1997), a widely known semistructured diagnostic interview which assesses 10 Axis II Personality Disorders from the DSM-IV (APA, 2000), and the Depressive and Passive-Aggressive Personality Disorders (included in DSM-IV's appendix).
  This assessment was carried out by researchers who had special training in the diagnosis of Personality Disorders and previous experience administering the SCID-II interview.

REFERENCES:
- [Derived] Gibbon S, Khalifa NR, Cheung NH, Vollm BA, McCarthy L. Psychological interventions for antisocial personality disorder. Cochrane Database Syst Rev. 2020 Sep 3;9(9):CD007668. doi: 10.1002/14651858.CD007668.pub3. PMID 32880104
- [Derived] Brazao N, Rijo D, Salvador MDC, Pinto-Gouveia J. The effects of the growing pro-social program on cognitive distortions and early maladaptive schemas over time in male prison inmates: A randomized controlled trial. J Consult Clin Psychol. 2017 Nov;85(11):1064-1079. doi: 10.1037/ccp0000247. PMID 29083222
- [Derived] Brazao N, Rijo D, Salvador MDC, Pinto-Gouveia J. Promoting emotion and behavior regulation in male prison inmates: A secondary data analysis from a randomized controlled trial testing the efficacy of the growing pro-social program. Law Hum Behav. 2018 Feb;42(1):57-70. doi: 10.1037/lhb0000267. Epub 2017 Oct 26. PMID 29072472